CLINICAL TRIAL: NCT00304213
Title: Does Testosterone Improve Function in Hypogonadal Older Men
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: Study never started, PI relocation
Sponsor: North Florida Foundation for Research and Education (Other)
Collaborators: Solvay Pharmaceuticals (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 79-06
Record Dates: First submitted 2006-03-16; First posted 2006-03-17 (Estimated); Last update posted 2015-02-13 (Estimated); Status verified 2015-02

CONDITIONS: Hypogonadism
Keywords: hypogonadism; testosterone; aging; Total testosterone < 300 ng/dL; Bioavailable testosterone < 70 ng/dL
MeSH Terms: conditions — Hypogonadism | interventions — Testosterone

INTERVENTIONS:
Drug: Testosterone

SUMMARY:
This is a randomized controlled trial of testosterone replacement therapy in hypogonadal men age > 60 years. The goal is to assess the safety and efficacy of TRT in men age > 60 years.

ELIGIBILITY:
Inclusion Criteria:

age 60-80 yrs serum total testosterone < 300 ng/dL serum bioavailable testosterone < 70 ng/dL

Exclusion Criteria:

unable to provide informed consent history of prostate or breast cancer untreated sleep apnea

Ages: 60 Years to 80 Years | Sex: Male
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2006-03; Study Completion 2009-04 (Estimated)

PRIMARY OUTCOMES:
Physical function
Cognitive function

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Mulligan, MD, Principal Investigator — Director, GRECC
Locations (1):
- Nf/Sg Vhs, Gainesville, Florida, United States